CLINICAL TRIAL: NCT00898547
Title: Additional Circulating Markers of Angiogenesis and Disease in Mesothelioma Patients Treated on CALGB 30107
Brief Title: Biomarkers of Angiogenesis and Disease in Patients With Unresectable Malignant Mesothelioma Treated on Clinical Trial CALGB-30107
Status: Terminated | Type: Observational
Why Stopped: Poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150509; U10CA031946 (NIH); CDR0000491313 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; recurrent malignant mesothelioma; epithelial mesothelioma; sarcomatous mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained from patients participating on CALGB-30107.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Serum samples previously obtained from patients on protocol CALGB-30107 are tested for levels of thrombospondin I serum, vascular endothelial growth factor receptor I, fibroblast growth factor, transforming growth factor, and mesothelin using enzyme-linked immunosorbent assays (ELISA).
  Interventions: Other: immunoenzyme technique; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about cancer and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at biomarkers of angiogenesis and disease in patients with unresectable malignant mesothelioma treated on clinical trial CALGB-30107.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if elevated levels of thrombospondin I serum levels, vascular endothelial growth factor receptor I, fibroblast growth factor, transforming growth factor, and mesothelin portend a poor prognosis in patients with unresectable malignant mesothelioma treated with vatalanib on protocol CALGB-30107.
* Determine if elevated levels of thrombospondin I serum levels, vascular endothelial growth factor receptor I, fibroblast growth factor, transforming growth factor, and mesothelin correlate with response or stable disease in these patients.

OUTLINE: Serum samples previously obtained from patients on protocol CALGB-30107 are tested for levels of thrombospondin I serum, vascular endothelial growth factor receptor I, fibroblast growth factor, transforming growth factor, and mesothelin using enzyme-linked immunosorbent assays (ELISA).

PROJECTED ACCRUAL: A total of 47 specimens will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignant mesothelioma

  * Unresectable disease
* Must have received treatment with vatalanib on protocol CALGB-30107

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously enrolled on CALGB-30107 diagnosed with malignant mesothelioma.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2005-11; Primary Completion 2006-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Level of biomarkers, including thrombospondin I, vascular endothelial growth factor receptor I, fibroblast growth factor, transforming growth factor, and mesothelin (high vs low) | baseline

SECONDARY OUTCOMES:
Effect of biomarker expression level on overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Kratzke, MD, Study Chair — Masonic Cancer Center, University of Minnesota